CLINICAL TRIAL: NCT01696591
Title: The Long-Term Safety and Efficacy Follow-up Study of Subjects Who Completed the Phase I Clinical Trial of Neurostem®-AD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Duk Lyul Na (Other)
Collaborators: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Duk Lyul Na, Professor of Neurology, Sungkyunkwan University School of Medicine, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: MP-CR-007-F/U
Record Dates: First submitted 2012-09-07; First posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Delirium, Dementia, Amnestic, Cognitive Disorders; Mental Disorders
Keywords: Alzheimer, Mesenchymal Stem Cells, Umbilical Cord Blood
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NEUROSTEM®-AD: A single administration of human umbilical cord blood-derived mesenchymal stem cells through a brain surgery
  DOSE A - 250,000 cells per entry site, 3 million cells per brain; DOSE B - 500,000 cells per entry site, 6 million cells per brain
  Interventions: Biological: NEUROSTEM®-AD
- Control Group: A group of subjects with comparable demographics (age and gender) and disease characteristics [Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB)] as the NEUROSTEM®-AD-treated group, but did not receive the treatment with NEUROSTEM®-AD and were continued on conventional therapy. Restrictions in the concurrent use of drug therapy are as follows:
  Patients are, in principle, permitted to continue the drug therapy they were on prior to the enrollment, for the treatment of concurrent illnesses other than Dementia, such as hypertension, diabetes mellitus, or hyperlipidemia.
  For drugs used in the treatment of dementia, behavior-modifying drugs can be added to the pharmacological regimen of a subject during the course of the study. However, adding a new cognitive enhancer, such as donepezil, memantine, galantamine, rivastigmine, is not permitted while dose adjustment is permitted given that the drug had been in use prior to the initiation of the study.

INTERVENTIONS:
Biological: NEUROSTEM®-AD — NEUROSTEM®-AD was administered to eligible subjects in the early part of the Phase I clinical study. In this follow-up study, no intervention will be performed.
  Other Names: human umbilical cord blood-derived mesenchymal stem cells (hUCB-MSCs)
  Groups: NEUROSTEM®-AD

SUMMARY:
The purpose of the study is to determine the long-term safety and exploratory efficacy of NEUROSTEM®-AD, administered via an open brain surgery to subjects with dementia of the Alzheimer's type, who were eligible for and enrolled in the earlier part of the phase I. Aside from the subjects who completed the earlier part of the Phase I, 3 additional subjects with comparable demographics and disease characteristics as the treatment group will be enrolled into a control group, followed-up for 3 months, and compared for various disease progression indicators with the treatment group.

The hypothesis is that NEUROSTEM®-AD is safe and effective in the treatment of dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
This is a long-term follow up study of the earlier part of the phase I, during which the safe and effective dose(safety) of NEUROSTEM®-AD was determined for implantation into the brains of subjects with Dementia of the Alzheimer's type. Subjects with Dementia of the Alzheimer's type, who signed the informed consent form and meet the eligibility criteria, were implanted with a single dose of NEUROSTEM®-AD, hUBC-MSCs, into the brain. The subjects were hospitalized for 5 to 10 days following the surgical implantation and were observed for acute adverse events: Gradient echo MRI within the the 24 hours post-op, vital signs, clinical laboratory tests, chest x-rays within Day 2. On Day 14, DLT was assessed, and the subjects were followed up on the safety and disease progression of dementia (of the Alzheimer's type) for 12 weeks post-implantation.

In this part of the study, the subjects described above will be followed-up for upto Month 24, and 3 additional subjects with comparable demographics and disease characteristics as the treatment group (refer to Inclusion/Exclusion Criteria) will be enrolled as a control group, followed up for 3 months and compared with the treatment group for various indicators of the disease progression.

ELIGIBILITY:
TEST GROUP

Inclusion Criteria:

* Subjects who have enrolled and completed the Phase I cliical trial: The Safety and The Efficacy Evaluation of NEUROSTEM®-AD in Patients With Alzheimer's Disease
* Subjects who are willing to participate in the study and sign the consent form

Exclusion Criteria:

* Females who are pregnant or nursing
* Subjects who have participated in another clinical study within the 3 months prior to the initiation of this study
* Subjects who are restricted from undergoing exams perfomed during the study (i.e. MRI, CT, or PET screening)
* Subjects who the principal investigator considers inappropriate for participation in the study due to any reasons other than those listed above

CONTROL GROUP

Inclusion Criteria:

* Patients with a moderate alzheimer's disease, diagnosed with a dementia of alzheimer's type, according to the DSM-VI and NINCDS-ADRDA criteria, and shows amyloid-positive in a PIB-PET

Exclusion Criteria:

* Subjects with a psychological disease (i.e. depression, schizophrenia, bipolar disorder, etc)
* Subjects with a dementia caused by other degenerative neurological diseases (infection of the CNS, such as HIV or Syphilis), head trauma, Creutzfeld-Jacob disease, Pick's disease, Huntington's disease, and Parkinson's disease)
* Subjects with a vascular dementia as determined by the clinical criteria of DSM IV and the imaging criteria of Erkinjuntii
* Subjects with severe white matter hyperintensities (WMH); Severe WMH is defined as, according to Clinical Research Center for Dementia of South Korea, a condition in which the deep white matter is 25 mm or greater and the periventricular capping/banding is 10 mm or greater in lengths.
* Subjects with a history of stroke within the 3 months prior to the study enrollment
* Subjects with a severe liver disease (ALT/AST values are higher than twice the normal range)
* Subjects with a severe renal disease (1.5mg/dL or more of serum creatinine)
* Pregnant or lactating women
* Subjects with abnormal findings of the clinical laboratory values at Visit 1:
* Hemoglobin < 9.5g/dL in male < 9.0 g/dL in female
* Total WBC count < 3000/mm3
* Total bilirubin ≥ 3 mg/dL
* Subjects with a suspected active lung disease, based on the chest X-ray result at Visit 1
* Females of childbearing age who does not practice medically acceptable method of contraception during the study
* Subjects who have previously failed Screening for participation in this study
* Subjects who have participated in another clinical study within the 3 months prior to the initiation of this study
* Subjects with a bleeding disorder (platelet count < 150,000/mm3; PT ≥ 1.5; INR or aPTT ≥ 1.5 X control
* Subjects with a cancer (including brain tumor)
* Subjects with a history of alcohol or drug abuse
* Subjects who are restricted from undergoing exams perfomed during the study (i.e. MRI, CT, or PET screening)
* Patients who the principal investigator considers inappropriate for participation in the study due to any reasons other than those listed above

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients, who were administered with NEUROSTEM®-AD in the earlier part of the Phase I study, will be compared with the patients, who have similar demographics and disease characteristics as the subjects in the test group but have not been treated with NEUROSTEM®-AD.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Safety | upto 24 months post-op
  Incidence rate ot adverse events (vital signs, physical examination, mixed lymphocyte reaction, and laboratory tests)

SECONDARY OUTCOMES:
Efficacy | upto 24 months post-op
  Primary Efficacy Variable:
  ADAS-cog response rate, ADAS-cog response is defined as when ADAS-cog score at the end of the study is not worse than the Baseline score.
  Secondary Efficacy Variables:
  * Changes in Seoul Instrumental Activities of Daily Living (S-IADL)
  * Changes in Mini Mental State Examination Korean verson (K-MMSE)
  * Changes in Caregiver-administered Neuropsuchiatric Inventory
  * Changes in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)
  * Changes in CMRglc: regional cerebral metabolic rate for glucose (FDG-PET)

CONTACTS AND LOCATIONS:
Overall Officials: Duk L. Na, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Seo SW, Chang JW, Lee JI, Kim CH, Chin J, Choi SJ, Kwon H, Yun HJ, Lee JM, Kim ST, Choe YS, Lee KH, Na DL. Stereotactic brain injection of human umbilical cord blood mesenchymal stem cells in patients with Alzheimer's disease dementia: A phase 1 clinical trial. Alzheimers Dement (N Y). 2015 Jul 26;1(2):95-102. doi: 10.1016/j.trci.2015.06.007. eCollection 2015 Sep. PMID 29854930
- See also: The Safety and The Efficacy Evaluation of NEUROSTEM®-AD in Patients With Alzheimer's Disease — http://clinicaltrials.gov/ct2/show/NCT01297218?term=neurostem&rank=1